CLINICAL TRIAL: NCT04549454
Title: Extension and Online Adaptation of the FITSTART Parent-based Intervention to Reduce Drinking Among First-year Students
Brief Title: Parent Feedback Intervention Targeting Student Transitions and Alcohol Related Trajectories (+) Efficacy Study
Acronym: FITSTART+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola Marymount University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Dr. Joseph LaBrie, Professor of Psychology, Loyola Marymount University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LoyolaMarymountU; R34AA026422 (NIH)
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Results first posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Alcohol Drinking; Alcohol Problem Drinking; Parenting
Keywords: Parent Intervention; Alcohol Intervention; College Student Drinking
MeSH Terms: conditions — Alcohol Drinking; Alcoholism; Alcohol Drinking in College

STUDY DESIGN:
Who Masked: Participant
Masking Description: Intervention condition is randomly assigned and the intervention delivery is digital, through a web app. Senior members of the research team will have a record of the participants randomized to each condition but the delivery of all intervention content is automated within the app. Junior members of the research team responsible for tracking participants and sending follow-up survey reminders will not be aware of participant condition assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention App (Experimental): Students in arm of the study will have a parent who has access to the following content in the parent app: (a) FITSTART+ PBI materials (personalized normative feedback quiz, information on college student drinking, and alcohol-specific advice for parents of first year students); (b) general advice for parents of college students (e.g., improving communication; reducing conflict); (c) information about university resources; and (d) a community section (parents can view other parent profiles, submit family photos, and view family photos submitted by other parents).
  Interventions: Behavioral: FITSTART+ PBI
- Control App (Placebo Comparator): Students in this arm of the study will have a parent who has access to the following content in the parent app: (a) general advice for parents of college students (e.g., improving communication; reducing conflict); (b) information about university resources; and (c) a community section (parents can view other parent profiles, submit family photos, and view family photos submitted by other parents).
  Interventions: Behavioral: General Parenting Advice

INTERVENTIONS:
Behavioral: FITSTART+ PBI — Personalized normative feedback on other parents behaviors + alcohol-specific parenting advice + general parenting advice
  Arms: Intervention App
Behavioral: General Parenting Advice — General parenting advice
  Arms: Control App

SUMMARY:
FITSTART (Feedback Intervention Targeting Student Transitions and Risk Trajectories) is a parent-based social norms intervention that has been shown to reduce risky drinking in incoming first year students.This program uses normative feedback to correct parents overestimation of other parents negative alcohol-related parenting practices (e.g., number of drinks parents would permit their college student to consume). Theory and research suggests that correcting those common misperceptions can motivate parents to adjust their own behaviors (e.g., reducing the number of drinks they would permit), which, in turn, can impact college student drinking. Despite FITSTARTs success, the design of the program limits participation to only students who have parents who can attend on-campus orientation sessions during the summer months before the start of the Fall semester. To address this limitation and extend the previous work, the proposed randomized clinical trial (RCT) will evaluate the efficacy of an online adaptation of the FITSTART(+) PBI program. To examine the efficacy of the newly developed FITSTART+ PBI web app, the proposed RCT will use a longitudinal design to examine if students self-report drinking and related negative consequences during their first semester in college significantly differed between FITSTART+ PBI (intervention app) and a control version of the app. Self-reported drinking and consequences are expected to be lower amongst students with parents randomized to FITSTART+ PBI relative to those with parents randomized to the control app.

DETAILED DESCRIPTION:
Heavy episodic drinking (HED) rates remains at unacceptably high levels on college campuses. Researchers on parent-based interventions (PBIs) has revealed promising results. but studies have generally failed to reduce HED in college students. FITSTART was developed to address two limitations of traditional PBIs that may contribute to the lack of the aforementioned effects: (I) they are purely informational and (II) they typically lack a motivational component to capture parents' attention and increase motivation to proactively engage their students. Pilot work has revealed that parents display predictable normative misperceptions (e.g., overestimate how approving other parents are of drinking and underestimate how often other parents engage with their students about drinking). As predicted by social norms theory, these false beliefs are associated with parents displaying more approving attitudes themselves and communicating less frequently. Correcting these norms should motivate parents to proactively engage their child in risk-reducing directions. FITSTART combined a social norms feedback component with informational material ("tips") characteristic of a traditional PBI in an in-person interactive format and successfully reduced HED. While the effects on weekly drinking, HED, and non-drinker alcohol use initiation were robust 1-month into college (3-months post intervention). FITSTART's usefulness as a universal approach is limited because it was delivered to parent groups on-campus during pre-college orientation sessions and many colleges do not hold summer orientations and/or lack the resources to administer FITSTART. To address this limitation, a web-based platform (or app) was developed using a new cutting-edge modality that draws from the computer science literature on virtual co-presence to create an online environment that mimics the effects of a live group social norms session.

The current pilot study seeks to evaluate the efficacy of the FITSTART+ PBI in a randomized control trial (RCT) by evaluating changes in incoming first-year students' alcohol use and related negative consequences during the transition into college. The sample will consist of traditional first year students (17-20 years of age) from Loyola Marymount University who completed consent and the baseline survey, and whose parents downloaded and registered for the FITSTART+ intervention or control app. Parents will be invited to download the intervention/control app two weeks prior to their student's arrival on campus in the fall (beginning of August). To examine the short- and long-term effects of the intervention, students will complete a baseline survey at the end of July (pre- matriculation) and two follow-up surveys, approximately 1 month (October) and 6 months (April) after the students arrive on campus in the spring.

ELIGIBILITY:
Inclusion Criteria:

First-year incoming LMU student consented to participate in the study and their parent/guardian created a profile on the app

Exclusion Criteria:

Outside of the students age range

Ages: 17 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 266 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph W LaBrie, PhD, Principal Investigator — Loyola Marymount University
Locations (1):
- Loyola Marymount, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Study results will be reported in aggregate, so that individual participants will not be identifiable in any research reports or presentations of the proposed study. A de-identified dataset will be made available to researchers 1 year after the initial publication of results. This dataset will include participant demographics and outcome measures assessed at baseline and the follow-up surveys. A data dictionary will be provided.
Supporting Information: Study Protocol, ICF
Time Frame: 1 year following publication of results.
Access Criteria: Study materials and data will be made available to the public on secure web portal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The university's admission's office emailed eligible first-year students an invite to take part in a 3-part longitudinal survey study (July 2021). Parents of students who completed the baseline survey were invited via email to join a free online program designed to help them support their student's college transition (Aug 2021). Invited parents were randomized to receive a web URL linking to either the intervention or control version of the program.
Period: T1 to T2
Arm/Group | Intervention App | Control App
Started (Note that the participant flow reported here reflects the period between the student baseline (July 2021 [T1]) and first follow-up (October 2021 [T2]) surveys. Thus, the number of participants reported during this period reflects the number of students who completed the surveys between T1 and T2. Students, not parents, are the ones who reported on outcomes. Parent data was not collected and therefore we could not include them in the Participant Flow.) | 134 | 132
Completed | 112 | 106
Not Completed | 22 | 26
Not completed — Lost to Follow-up | 22 | 26
Period: T1 to T3
Arm/Group | Intervention App | Control App
Started (Note that the participant flow reported here reflects the period between the student baseline (July 2021 [T1]) and second follow-up (February 2022 [T3]) surveys. Thus, the number of participants reported during this period reflects the number of students who completed the surveys between T1 and T3. Students, not parents, are the ones who reported on outcomes. Parent data was not collected and therefore we could not include them in the Participant Flow.) | 134 | 132
Completed | 103 | 96
Not Completed | 31 | 36
Not completed — Lost to Follow-up | 31 | 36

BASELINE CHARACTERISTICS:
Population: Baseline data was only collected for students because all outcomes for this trial are student behaviors. Thus, the participant attributes are those of the students and not their parents. Additionally, there are some discrepancies between the number of participants indicated in the Participant Flow and the number of participants who reported on outcomes. This is due to some participants not providing answers on some survey questions (i.e., survey questions were not forced response).
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention App | Control App | Total
Number analyzed (Participants) | 134 | 132 | 266
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 129 | 124 | 253
  Between 18 and 65 years | 5 | 8 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.91 (0.40) | 17.91 (0.45) | 17.91 (0.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 75 | 154
  Male | 55 | 57 | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 34 | 66
  Not Hispanic or Latino | 102 | 98 | 200
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 17 | 15 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 16 | 30
  White | 69 | 72 | 141
  More than one race | 32 | 25 | 57
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 134 | 132 | 266
Typical Weekly Drinking [Mean (Standard Deviation); unit: Typical alcohol drinks consumed per week] — Participants reported the typical quantity of standard alcohol drinks consumed on each day of the week during the past 30 days using the Daily Drinking Questionnaire. Quantity of drinks reported on each day of the week were then summed to create a composite variable assessing typical weekly drinking.
  Typical alcohol drinks consumed per week | 1.97 (3.70) | 1.98 (3.78) | 1.97 (3.74)
Consequences [Mean (Standard Deviation); unit: Types of alcohol consequences] — The number of types of negative alcohol-related consequences experienced out of a list of 14 common negative alcohol-related consequences in the past month were summed to create a composite variable for consequences.
  Types of alcohol consequences | 1.34 (1.96) | 1.35 (2.04) | 1.34 (2.00)
Quantity/Frequency/Peak Alcohol Use [Mean (Standard Deviation); unit: Peak alcoholic beverages consumed] — An item assessing the number of maximum drinks on one occasion from the Frequency, Quantity, Max (FQM) measure was used to assess peak drinks on one occasion over the past 30 days.
  Peak alcoholic beverages consumed | 1.78 (2.53) | 2.17 (3.16) | 1.97 (2.86)
HED [Mean (Standard Deviation); unit: HED events] — An item assessing the number of times students reported a heavy episodic drinking (HED) event in the past two weeks.
  HED events | 0.42 (1.05) | 0.56 (1.44) | 0.49 (1.26)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Typical Weekly Drinking at 1 Month
Description: At baseline and the 1-month follow-up, participants reported the typical quantity of standard alcohol drinks consumed on each day of the week during the past 30 days using the Daily Drinking Questionnaire. Quantity of drinks reported on each day of the week at baseline and 1-month were then summed (separately) to create a composite variable assessing typical weekly drinking at each time point. To compute the outcome, the 1-month measure of typical drinks per week was subtracted from the baseline measure of typical drinks per week such that a positive value indicates a decrease in consumption during this period and a negative value indicates an increase in consumption during this period.
Time Frame: baseline, 1 month
Measure: Mean (Standard Deviation); unit: typical alcohol drinks consumed per week
Arm/Group | Intervention App | Control App
Number analyzed (Participants) | 111 | 106
typical alcohol drinks consumed per week | 1.67 (3.65) | 1.82 (3.77)
Statistical Analysis 1: Comparison: Intervention App vs Control App; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, in examining Time*Arm interactions on weekly drinks. To probe the significant Time*Arm interaction, a Tukey post-hoc test examined the change in weekly drinks from baseline to the 1-month follow-up in the Intervention Arm versus the Control Arm; Test type: Superiority; p = .985, Tukey-Kramer; Mean Difference (Final Values) = -0.011, Standard Error of Mean 0.598

2. Primary Outcome: Change From Baseline Typical Weekly Drinking at 6 Months
Description: At baseline and the 6-month follow-up, participants reported the typical quantity of standard alcohol drinks consumed on each day of the week during the past 30 days using the Daily Drinking Questionnaire. Quantity of drinks reported on each day of the week at baseline and 1-month were then summed (separately) to create a composite variable assessing typical weekly drinking at each time point. To compute the outcome, the 6-month measure of typical drinks per week was subtracted from the baseline measure of typical drinks per week such that a positive value indicates a decrease in consumption during this period and a negative value indicates an increase in consumption during this period.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: typical alcohol drinks consumed per week
Arm/Group | Intervention App | Control App
Number analyzed (Participants) | 103 | 94
typical alcohol drinks consumed per week | 2.31 (5.20) | 2.21 (4.44)
Statistical Analysis 1: Comparison: Intervention App vs Control App; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, in examining Time*Arm interactions on weekly drinks. To probe the significant Time*Arm interaction, a Tukey post-hoc test examined the change in weekly drinks from baseline to the 6-month follow-up in the Intervention Arm versus the Control Arm; Test type: Superiority; p = .694, Tukey-Kramer; Mean Difference (Final Values) = 0.244, Standard Error of Mean 0.618

3. Primary Outcome: Change From Baseline Frequency of Alcohol Consequences at 1 Month
Description: At baseline and the 1-month follow-up, the number of types of negative alcohol-related consequences experienced out of a list of 14 common negative alcohol-related consequences (past 30 days) were summed to create a composite variable at each time point. To compute the outcome, the 1-month measure of negative consequences was subtracted from the baseline measure of negative consequences such that a positive value indicates a decrease in consequences during this period and a negative value indicates an increase in consequences during this period.
Time Frame: baseline, 1 month
Measure: Mean (Standard Deviation); unit: types of alcohol consequences
Arm/Group | Intervention App | Control App
Number analyzed (Participants) | 112 | 105
types of alcohol consequences | 0.24 (1.71) | 0.28 (2.22)
Statistical Analysis 1: Comparison: Intervention App vs Control App; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, in examining Time*Arm interactions on consequences. To probe the significant Time*Arm interaction, a Tukey post-hoc test examined the change in consequences from baseline to the 1-month follow-up in the Intervention Arm versus the Control Arm; Test type: Superiority; p = .889, Tukey-Kramer; Mean Difference (Final Values) = -0.045, Standard Error of Mean 0.327

4. Primary Outcome: Change From Baseline Frequency of Alcohol Consequences at 6 Months
Description: At baseline and the 6-month follow-up, the number of types of negative alcohol-related consequences experienced out of a list of 14 common negative alcohol-related consequences (past 30 days) were summed to create a composite variable at each time point. To compute the outcome, the 6-month measure of negative consequences was subtracted from the baseline measure of negative consequences such that a positive value indicates a decrease in consequences during this period and a negative value indicates an increase in consequences during this period.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: types of alcohol consequences
Arm/Group | Intervention App | Control App
Number analyzed (Participants) | 103 | 96
types of alcohol consequences | .52 (2.84) | .73 (3.30)
Statistical Analysis 1: Comparison: Intervention App vs Control App; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, in examining Time*Arm interactions on consequences. To probe the significant Time*Arm interaction, a Tukey post-hoc test examined the change in consequences from baseline to the 6-month follow-up in the Intervention Arm versus the Control Arm; Test type: Superiority; p = .582, Tukey-Kramer; Mean Difference (Final Values) = -0.186, Standard Error of Mean 0.338

5. Primary Outcome: Change From Baseline Quantity/Frequency/Peak Alcohol Use at 1 Month
Description: At baseline and the 1-month follow-up, an item assessing the number of maximum drinks on one occasion from the Frequency, Quantity, Max (FQM) measure was used to assess peak drinks on one occasion over the past 30 days. To compute the outcome, the 1-month measure of peak drinks was subtracted from the baseline measure of peak drinks such that a positive value indicates a decrease in consumption during this period and a negative value indicates an increase in consumption during this period.
Time Frame: baseline, 1 month
Measure: Mean (Standard Deviation); unit: Peak alcoholic beverages consumed
Arm/Group | Intervention App | Control App
Number analyzed (Participants) | 111 | 106
Peak alcoholic beverages consumed | .91 (2.46) | .98 (2.63)
Statistical Analysis 1: Comparison: Intervention App vs Control App; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, in examining Time*Arm interactions on peak drinks. To probe the significant Time*Arm interaction, a Tukey post-hoc test examined the change in peak drinks from baseline to the 1-month follow-up in the Intervention Arm versus the Control Arm; Test type: Superiority; p = .523, Tukey-Kramer; Mean Difference (Final Values) = -0.265, Standard Error of Mean 0.414

6. Primary Outcome: Change From Baseline Quantity/Frequency/Peak Alcohol Use at 6 Months
Description: At baseline and the 6-month follow-up, an item assessing the number of maximum drinks on one occasion from the Frequency, Quantity, Max (FQM) measure was used to assess peak drinks on one occasion over the past 30 days. To compute the outcome, the 6-month measure of peak drinks was subtracted from the baseline measure of peak drinks such that a positive value indicates a decrease in consumption during this period and a negative value indicates an increase in consumption during this period.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: Peak alcoholic beverages consumed
Arm/Group | Intervention App | Control App
Number analyzed (Participants) | 103 | 95
Peak alcoholic beverages consumed | 1.54 (3.43) | 1.36 (3.25)
Statistical Analysis 1: Comparison: Intervention App vs Control App; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, in examining Time*Arm interactions on peak drinks. To probe the significant Time*Arm interaction, a Tukey post-hoc test examined the change in peak drinks from baseline to the 6-month follow-up in the Intervention Arm versus the Control Arm; Test type: Superiority; p = .981, Tukey-Kramer; Mean Difference (Final Values) = 0.010, Standard Error of Mean 0.427

7. Primary Outcome: Change From Baseline Heavy Episodic Drinking at 1 Month
Description: At baseline and the 1-month follow-up, an item assessing the number of times students reported a heavy episodic drinking (HED) event in the past two weeks. To compute the outcome, the 1-month measure of HED was subtracted from the baseline measure of HED such that a positive value indicates a decrease in HED events during this period and a negative value indicates an increase in HED events during this period.
Time Frame: baseline, 1 month
Measure: Mean (Standard Deviation); unit: HED events
Arm/Group | Intervention App | Control App
Number analyzed (Participants) | 111 | 106
HED events | .41 (1.27) | .47 (1.44)
Statistical Analysis 1: Comparison: Intervention App vs Control App; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, in examining Time*Arm interactions on HED. To probe the significant Time*Arm interaction, a Tukey post-hoc test examined the change in HED from baseline to the 1-month follow-up in the Intervention Arm versus the Control Arm; Test type: Superiority; p = .889, Tukey-Kramer; Median Difference (Final Values) = -0.045, Standard Error of Mean 0.327

8. Primary Outcome: Change From Baseline Heavy Episodic Drinking at 6 Months
Description: as for outcome 7
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: HED events
Arm/Group | Intervention App | Control App
Number analyzed (Participants) | 103 | 96
HED events | .67 (1.67) | .56 (1.50)
Statistical Analysis 1: Comparison: Intervention App vs Control App; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, in examining Time*Arm interactions on HED. To probe the significant Time*Arm interaction, a Tukey post-hoc test examined the change in HED from baseline to the 6-month follow-up in the Intervention Arm versus the Control Arm; Test type: Superiority; p = .582, Tukey-Kramer; Mean Difference (Final Values) = -0.186, Standard Error of Mean 0.338

ADVERSE EVENTS:
Time Frame: Survey participants (students) were provided with phone and email at the start of each survey and encouraged to report any adverse events. The period to report adverse events for these participants was between the start of the T1 survey (baseline) and the end of the T3 (second follow-up) surveys. This period was approximately 8 months.
Arm/Group | Intervention App | Control App
All-Cause Mortality (participants affected / at risk) | 0/134 | 0/132
Serious Adverse Events (participants affected / at risk) | 0/134 | 0/132
Other Adverse Events (participants affected / at risk) | 0/134 | 0/132

LIMITATIONS AND CAVEATS:
This trial was conducted in the first on-campus semester post-Covid, and there were several restrictions regarding student life in effect. This likely affected student alcohol use by limiting social drinking events and willingness to engage in those events (depressing the levels of risky drinking). Thus, the ability to detect changes in drinking was likely to have been impacted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT04549454/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT04549454/SAP_001.pdf
  • Informed Consent Form (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT04549454/ICF_002.pdf